CLINICAL TRIAL: NCT06631274
Title: IVY: Intervention for Victimized Youth
Brief Title: Intervention for Victimized Youth
Acronym: IVY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, Lyndsay Jenkins, Principal Investigator, Florida State University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00004121; 1R21HD112660 (NIH)
Record Dates: First submitted 2024-10-04; First posted 2024-10-08 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Victimization
Keywords: peer victimization; bullying; trauma
MeSH Terms: conditions — Bullying; Wounds and Injuries | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: We are using a waitlist control model where half of the participants will be randomly assigned to the treatment condition. When that intervention is completed, the treatment will be offered to the waitlist participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 8 weeks of group counseling delivered in virtual environment (Other): The treatment to be piloted is a 8 week virtual group counseling intervention with a focus on teaching participants skills to overcome emotional difficulties (Visit 1-4) and avoiding re-victimization (Visit 5-Visit 8).
  Interventions: Behavioral: counseling
- control group (No Intervention): Participants in this arm do not receive the intervention at the same time as the treatment group.

INTERVENTIONS:
Behavioral: counseling — The intervention (IVY; Intervention for Victimized Youth) is an 8 week group counseling intervention delivered in a virtual environment.
  Arms: 8 weeks of group counseling delivered in virtual environment

SUMMARY:
IVY (Intervention for Victimized Youth). Just as ivy plants are strong and can flourish in difficult environments, the goal of IVY will be for targets of peer victimization to thrive academically and socially despite challenging circumstances.

DETAILED DESCRIPTION:
The project involves the development of a virtual intervention program for targets of peer victimization. Intervention for Victimized Youth (IVY) will improve upon many limitations of existing interventions described above since it is the first intervention program to specifically address the needs of targets of peer victimization from a trauma perspective. Moreover, it addresses key limitations of CBITS and increases the flexibility of the intervention by using a virtual delivery model. Just as ivy plants are strong and can flourish in difficult environments, the goal of IVY is for victimized youth to thrive academically and socially despite challenging circumstances. IVY uses a cognitive behavioral therapy (CBT) approach to address current distress due to peer victimization and teach strategies for handling any future peer victimization. Common elements of effective CBT-based trauma treatments are psychoeducation, emotion regulation skills, imaginal or in vivo exposure, cognitive processing, and/or problem solving. Several methods are used within sessions to teach the content, including psychoeducation, didactic teaching, modeling, role playing, and guided self-reflection.

The proposed 8-week intervention. The focus of the first 4 sessions will be on teaching skills to help students overcome emotional difficulties associated with being victimized. Weekly topics include: 1) Introduction & Psychoeducation, 2) Emotional Regulation Skill Building and Practice, 3) Identifying & Coping with Difficult Thoughts and Emotions, and 4) Connecting Thoughts, Emotions, and Behaviors. The last 4 sessions are specific to peer victimization issues with a focus on avoiding re-victimization since victimized youth often are victimized repeatedly and report that they defend other victims. Weekly topics include: 5) Options for Protecting Yourself, 6) Social Problem-Solving Skills, 7) Adaptive Thinking, and 8) Future Planning & Celebration. Participants will be taught several options for intervening. A decision-making process for evaluating social situations will be taught. Based on the outcome of that decision-making process, participants will be taught options for responding with the goal of avoiding re-victimized.

ELIGIBILITY:
Inclusion Criteria:

* current middle school student in US (defined as grades 6, 7, or 8)
* experience at least one instance of peer victimization in past month
* Have elevated or extremely elevated social-emotional distress score, as measured by the BESS (Behavior and Emotional Screening System)

Exclusion Criteria:

* not current middle school student
* not experience victimization in past month
* no elevated score on BESS

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Florida State University Department of Educational Psychology and Learning Systems, Tallahassee, Florida
  - Florida State University, Tallahassee, Florida

IPD SHARING:
Plan to Share IPD: No
Pilot program, unable to support requests for IPD

REFERENCES:
- See also: webpage about IVY — https://cehhs.fsu.edu/ivy

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited participants from September 2024 to March 2025. We sent out recruitment information to schools to share with families, conducted targeted online recruitment, posted physical flyers, and used word of mouth snowball recruitment strategies.
Pre-assignment Details: Parents initially completed an interest survey. Each response was evaluated to assess whether the child met the inclusion criteria and whether the response passed the validity checks to ensure it was not a bot. After passing these checks, a "pre-survey" was sent with a request for the child to complete assent and confirm they experienced at least one instance of bullying in the past month. After returning the second survey, they were randomly assigned to the treatment or control group.
Period: Overall Study
Arm/Group | 8 weeks of group counseling delivered in virtual environment | control group
Started | 23 | 25
Completed | 22 | 20
Not Completed | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 8 Weeks of Group Counseling Delivered in Virtual Environment | Control Group | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 22 | 20 | 42
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 12 | 17
  Male | 17 | 8 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 0 | 7
  Not Hispanic or Latino | 15 | 20 | 35
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 8 | 14
  White | 16 | 8 | 24
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Change in Social-emotional Distress
Description: The Behavioral and Emotional Screening System is a 30 item measure. For each item, participants decide how often a statement is true for them and respond using a 4-point Likert scale (0=never to 3=always). Personal adjustment is measured by 8 items (possible mean scores ranging from 0 to 3) and internalizing problems is measured by 10 items (possible mean scores ranging from 0 to 3). Mean item scores are computed for personal adjustment and internalizing problems, respectively, at pretest (time 1) and posttest (time 2). For both subscales, higher scores indicate greater difficulties, i.e., worse adjustment and worse internalizing issues.
Time Frame: Visit 1 (baseline); Visit 8 (8 weeks after baseline at the termination visit)
Measure: Mean (Standard Deviation); unit: mean item score on a scale
Arm/Group | 8 weeks of group counseling delivered in virtual environment | control group
Number analyzed (Participants) | 22 | 20
mean item score on a scale
  Personal adjustment at time 1 | 1.09 (0.53) | 1.07 (0.55)
  Personal adjustment at time 2 | 0.97 (0.61) | 1.00 (0.61)
  Internalizing Problems at time 1 | 1.16 (0.67) | 1.31 (0.56)
  Internalizing Problems at time 2 | 1.28 (0.55) | 1.24 (0.61)
Statistical Analysis 1: Comparison: 8 weeks of group counseling delivered in virtual environment vs control group; The outcome measure is personal adjustment; Test type: Equivalence — A one-way repeated measures ANOVA was conducted to examine the impact of intervention, in which participation in the intervention (treatment vs. control) was used as the between-subject factor and time points (time 1 and time 2) was used as the within-subject factor. The interaction between group and time was the focus and was reported; p = 0.646, ANOVA; one-way repeated measures ANOVA was conducted for personal adjustment; Mean Difference (Final Values) = -0.056, 95% CI 2-sided [-0.296 to 0.184] — Hedges' g=-0.14. The mean difference between the two time points (change) was computed as time2 minus time1. Hedges' g was the standardized mean difference between change in the treatment group and change in the control group
Statistical Analysis 2: Comparison: 8 weeks of group counseling delivered in virtual environment vs control group; The outcome measure is internalizing problems; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.196, ANOVA; one-way repeated measures ANOVA was conducted for internalizing problems; Mean Difference (Final Values) = 0.188, 95% CI 2-sided [-0.096 to 0.473] — Hedges' g=0.40. The mean difference between the two time points (change) was computed as time2 minus time1. Hedges' g was the standardized mean difference between change in the treatment group and change in the control group

2. Primary Outcome: Change in Knowledge of Self-protection Skills
Description: The Knowledge of Self-Protection Options (KSPO) scale consists of 9 items assessing the degree to which participants have knowledge of how to protect themselves. Participants are asked "If I am being bullied, I know how to..." then rate each item on a 3 point scale ranging from 0 (No), 1 (A little bit), or 2 (Yes). Mean scores were calculated for each participant, which could range from 0 to 2, which higher scores representing greater knowledge of how to protect oneself.
Time Frame: Visit 1 (baseline); Visit 8 (8 weeks after baseline at the termination visit)
Measure: Mean (Standard Deviation); unit: mean item score on a scale
Arm/Group | 8 weeks of group counseling delivered in virtual environment | control group
Number analyzed (Participants) | 22 | 20
mean item score on a scale
  Knowledge of Self-Protection Options at Time 1 | 1.18 (0.39) | 1.16 (0.41)
  Knowledge of Self-Protection Options at Time 2 | 1.59 (0.40) | 1.24 (0.37)
Statistical Analysis 1: Comparison: 8 weeks of group counseling delivered in virtual environment vs control group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.01, ANOVA; one-way repeated ANOVA was conducted; Mean Difference (Final Values) = 0.326, 95% CI 2-sided [0.112 to 0.539] — Hedges' g=0.92. The mean difference between the two time points (change) was computed as time2 minus time1. Hedges' g was the standardized mean difference between change in the treatment group and change in the control group

3. Primary Outcome: Change in Self-efficacy for Protecting Self
Description: The Self-Efficacy for Protecting Self (SEPS) scale consists of 8 items with the stem of "How do you rate your ability to engage in each action?" Response options range from 1 (I can not do this well at all) to 4 (I can do this very well). Mean scores were calculated for each participant, which could range from 1 to 4, which higher scores representing greater efficacy in protecting oneself.
Time Frame: Visit 1 (baseline); Visit 8 (8 weeks after baseline at the termination visit)
Population: For this measure, two participants selected the same response option for every item on the scale (e.g., selected "1" for every question, even validity items). We questioned the validity of their responses so we removed those two participants from the analysis for this outcome variable.
Measure: Mean (Standard Deviation); unit: mean item score on a scale
Arm/Group | 8 weeks of group counseling delivered in virtual environment | control group
Number analyzed (Participants) | 20 | 20
mean item score on a scale
  Self-Efficacy for Protecting Self at Time 1 | 4.52 (1.27) | 4.14 (1.23)
  Self-Efficacy for Protecting Self at Time 2 | 4.19 (1.26) | 5.19 (1.62)
Statistical Analysis 1: Comparison: 8 weeks of group counseling delivered in virtual environment vs control group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.11, ANOVA; one-way repeated measures ANOVA was conducted; Mean Difference (Final Values) = 0.681, 95% CI 2-sided [-0.187 to 1.549] — Hedges' g=0.51. The mean difference between the two time points (change) was computed as time2 minus time1. Hedges' g was the standardized mean difference between change in the treatment group and change in the control group

4. Primary Outcome: Change in Knowledge of Coping Skills
Description: Coping skills will be measured using the Brief COPE, which is a 28-item scale that assesses coping strategies. Items are rated on a scale from 1 (I haven't been doing this at all) to 4 (I've been doing this a lot). Avoidance coping is measured by 11 items and approach coping is measured by 12 items. Mean scores were calculated for each participant, which could range from 1 to 4, which higher scores representing greater knowledge of how to protect oneself.
Time Frame: Visit 1 (baseline); Visit 8 (8 weeks after baseline at the termination visit)
Measure: Mean (Standard Deviation); unit: mean item score on a scale
Arm/Group | 8 weeks of group counseling delivered in virtual environment | control group
Number analyzed (Participants) | 22 | 20
mean item score on a scale
  Avoidance coping at time 1 | 2.00 (0.46) | 2.17 (0.45)
  Avoidance coping at time 2 | 2.18 (0.41) | 2.08 (0.52)
  Approach coping at time 1 | 2.44 (0.56) | 2.56 (0.59)
  Approach coping at time 2 | 2.42 (0.58) | 2.86 (0.65)
Statistical Analysis 1: Comparison: 8 weeks of group counseling delivered in virtual environment vs control group; The outcome measure is avoidance coping; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.599, ANOVA; one-way repeated measures ANOVA was conducted for avoidance coping; Mean Difference (Final Values) = 0.078, 95% CI 2-sided [-0.212 to 0.367] — Hedges' g=0.16. The mean difference between the two time points (change) was computed as time2 minus time1. Hedges' g was the standardized mean difference between change in the treatment group and change in the control group
Statistical Analysis 2: Comparison: 8 weeks of group counseling delivered in virtual environment vs control group; The outcome measure is approach coping; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.044, ANOVA; one-way repeated measures ANOVA was conducted for approach coping; Mean Difference (Final Values) = 0.316, 95% CI 2-sided [0.152 to 0.617] — Hedges' g=0.63. The mean difference between the two time points (change) was computed as time2 minus time1. Hedges' g was the standardized mean difference between change in the treatment group and change in the control group

5. Secondary Outcome: Change in Peer Victimization
Description: The victim subscale of the Bullying Participant Behavior Questionnaire will be used to assess traditional/in-person victimization. The scale consists of 10 items Participants respond ranging from 1 (never) to 5 (7 or more times) in the past 30 days. A mean score was calculated for each participant, which could range from 1 to 5 with higher scores representing more victimization.
Time Frame: Visit 1 (baseline); Visit 8 (8 weeks after baseline at the termination visit)
Measure: Mean (Standard Deviation); unit: mean item score on a scale
Arm/Group | 8 weeks of group counseling delivered in virtual environment | control group
Number analyzed (Participants) | 22 | 20
mean item score on a scale
  Peer victimization at time 1 | 2.60 (1.22) | 2.69 (1.10)
  Peer victimization at time 2 | 2.55 (1.11) | 1.63 (0.83)
Statistical Analysis 1: Comparison: 8 weeks of group counseling delivered in virtual environment vs control group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p < .01, ANOVA; one-way repeated measures ANOVA was conducted; Mean Difference (Final Values) = 1.024, 95% CI 2-sided [0.284 to 1.764] — Hedges' g=0.85. The mean difference between the two time points (change) was computed as time2 minus time1. Hedges' g was the standardized mean difference between change in the treatment group and change in the control group

6. Secondary Outcome: Change in Cyber Victimization
Description: The victim subscale of the Cyber Bullying Participant Rating Scales will be used to assess cyber victimization. The scale consists of 11 items. The 6-point Likert scale (1 = not at all to 6 = many times a week) requires participants to rate how often they have been a victim. A mean score was calculated for each participant, which could range from 1 to 6 with higher scores representing more cyber victimization.
Time Frame: Visit 1 (baseline); Visit 8 (8 weeks after baseline at the termination visit)
Measure: Mean (Standard Deviation); unit: mean item score on a scale
Arm/Group | 8 weeks of group counseling delivered in virtual environment | control group
Number analyzed (Participants) | 22 | 20
mean item score on a scale
  Cyber victimization at time 1 | 1.47 (0.68) | 1.39 (0.66)
  Cyber victimization at time 2 | 2.18 (1.06) | 1.67 (0.82)
Statistical Analysis 1: Comparison: 8 weeks of group counseling delivered in virtual environment vs control group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0498, ANOVA; one-way repeated measures ANOVA was conducted; Mean Difference (Final Values) = -0.589, 95% CI 2-sided [-1.178 to -0.0005] — Hedges' g=-0.61. The mean difference between the two time points (change) was computed as time2 minus time1. Hedges' g was the standardized mean difference between change in the treatment group and change in the control group

7. Secondary Outcome: Change in Traumatic Stress Symptoms
Description: Child PTSD Symptom Screener-Self-Report Version for DSM-5 will be used to assess traumatic stress symptoms. The scale consists of 16 self-report items with item responses ranging from 0 (not at all) to 4 (6 or more times a week/almost always). A mean score was calculated for each participant, which could range from 0 to 4 with higher scores representing more traumatic stress.
Time Frame: Visit 1 (baseline); Visit 8 (8 weeks after baseline at the termination visit)
Measure: Mean (Standard Deviation); unit: mean item score on a scale
Arm/Group | 8 weeks of group counseling delivered in virtual environment | control group
Number analyzed (Participants) | 22 | 20
mean item score on a scale
  Traumatic stress at time 1 | 2.11 (0.68) | 2.31 (0.74)
  Traumatic stress at time 2 | 2.15 (0.73) | 2.22 (0.56)
Statistical Analysis 1: Comparison: 8 weeks of group counseling delivered in virtual environment vs control group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.182, ANOVA; one-way repeated measures ANOVA was conducted; Mean Difference (Final Values) = 0.261, 95% CI 2-sided [-0.127 to 0.650] — Hedges' g=0.41. The mean difference between the two time points (change) was computed as time2 minus time1. Hedges' g was the standardized mean difference between change in the treatment group and change in the control group

8. Secondary Outcome: Change in Social Support
Description: The Child and Adolescent Social Support Scale will be used to assess perceptions of social support. Only the peer support scale will be used. It consists of 12 items with response options ranging from 1 (never) to 6 (always). A mean score was calculated for each participant, which could range from 1 to 6 with higher scores representing more social support.
Time Frame: Visit 1 (baseline); Visit 8 (8 weeks after baseline at the termination visit)
Population: Due to an error in the online survey, some participants did not complete the full social support scale, therefore there was missing data on this outcome variable. Participants who did not respond to at least 50% of the items were excluded from analysis.
Measure: Mean (Standard Deviation); unit: mean item score on a scale
Arm/Group | 8 weeks of group counseling delivered in virtual environment | control group
Number analyzed (Participants) | 14 | 9
mean item score on a scale
  Peer support at time 1 | 3.96 (1.10) | 4.05 (1.15)
  Peer support at time 2 | 4.02 (0.89) | 4.15 (1.20)
Statistical Analysis 1: Comparison: 8 weeks of group counseling delivered in virtual environment vs control group; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.927, ANOVA; one-way repeated measures ANOVA was conducted; Mean Difference (Final Values) = -0.030, 95% CI 2-sided [-0.612 to 0.551] — Hedges' g=-0.04. The mean difference between the two time points (change) was computed as time2 minus time1. Hedges' g was the standardized mean difference between change in the treatment group and change in the control group

ADVERSE EVENTS:
Time Frame: Data were collected over a 10 week period, with Time 1 data collected the week before the intervention began and Time 2 data collected during the week week after the intervention ended. The intervention was 8 weekly sessions.
Description: No different from clinicaltrial.gov definition
Arm/Group | 8 weeks of group counseling delivered in virtual environment | control group
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/22 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-10-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT06631274/Prot_001.pdf
  • Statistical Analysis Plan (2024-10-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT06631274/SAP_002.pdf
  • Informed Consent Form (2024-10-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT06631274/ICF_000.pdf